CLINICAL TRIAL: NCT00632385
Title: An Open-label Study of Eletriptan for the Acute Treatment of Migraine in Migraine Sufferers Who Are Dissatisfied With Rizatriptan Therapy
Brief Title: Efficacy and Safety of Eletriptan for the Treatment of Migraine in Patients Not Satisfied With Rizatriptan Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1601092
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eletriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Eletriptan

INTERVENTIONS:
Drug: Eletriptan — 40 mg oral tablet for migraine attack, followed by 40 mg oral tablet if migraine reoccurred >2 hours from first dose and within 24 hours of first dose

SUMMARY:
To assess the efficacy and safety of eletriptan for migraine headaches in subjects who were not satisfied with rizatriptan therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine headache according to International Headache Society criteria and migraine headaches for at least 1 year
* Eletriptan naive
* Previously treated with rizatriptan and failed to achieve a satisfactory response within the past 12 months

Exclusion Criteria:

* Non-migraine headaches on average more than 6 days per month or have less than 24 hours of freedom from headache between migraine attacks
* Migraine attacks that are atypical or chronic daily headaches
* A history of migraine with prolonged aura, familial hemiplegic migraine, basilar migraine, migrainous infarction, migraine aura without headache, migraine with acute onset aura

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2003-01; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in headache pain severity | 1, 2, 4, and 24 hours

SECONDARY OUTCOMES:
Functional impairment | 1, 2, 4, and 24 hours
Work Productivity Questionnaire | Week 10
Time Loss | Week 10
Subject Preference Questionnaire | Week 10
Global Evaluation | Week 10
Subject Satisfaction Scale | Week 10
Associated Symptoms | 1, 2, 4, and 24 hours
Use of Rescue Medication | Week 10
Adverse events | Week 10
Vital signs | Week 10
Physical examination | Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Alexandria, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601092&StudyName=Efficacy%20and%20Safety%20of%20Eletriptan%20for%20the%20Treatment%20of%20Migraine%20in%20Patients%20Not%20Satisfied%20with%20Rizatriptan%20Therapy